CLINICAL TRIAL: NCT05556395
Title: Global Blood-Brain Barrier Disruption and Post-Stroke Cognitive Decline
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00312030
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Ischemic Stroke
Keywords: blood-brain barrier; post-stroke cognitive impairment and dementia; vascular cognitive impairment and dementia; Alzheimer's disease and related dementias; stroke
MeSH Terms: conditions — Ischemic Stroke; Dementia; Alzheimer Disease; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to gain a better understanding of why some individuals who have suffered a stroke experience post-stroke cognitive decline. Specifically this study is testing whether global disruption of the blood-brain barrier detected at the time of the stroke is informative about the risk of post-stroke cognitive decline over the next 3 years.

DETAILED DESCRIPTION:
It is well known that ischemic stroke is a risk factor for developing dementia. Prior studies have shown that after a stroke, there can be a change in the trajectory of cognitive performance with acceleration of decline. The mechanism of this phenomenon has not been established. It is known that vascular changes in the brain, referred to as cerebral small vessel disease, are associated with cognitive decline and dementia. Cerebral small vessel disease is readily seen on MRI scans of the brain, and the larger the burden of these findings, the higher the risk of cognitive deficits. Disruption of the blood-brain barrier has been implicated in the development of the changes seen on MRI. Acute stroke has been shown to disrupt the blood-brain barrier, even in parts of the brain not directly affect by the stroke. The investigators hypothesize that when there is diffuse blood-brain barrier disruption in response to an acute stroke it sets off a cascade of changes in the brain that lead to post-stroke cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke demonstrated on an MRI scan that includes perfusion imaging with an exogenous contrast agent

Exclusion Criteria:

* Inability to perform telephone-based cognitive assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are admitted to the hospital and diagnosed with an ischemic stroke based on an MRI scan that also includes perfusion imaging with an exogenous contrast agent and are will/able to be contacted for serial phone-based cognitive evaluations.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in Cognition (Cognitive Decline) | Assessments occur every 6 months for 3 years
  Serial telephone-based cognitive assessments will be performed to detect cognitive changes (cognitive decline).

CONTACTS AND LOCATIONS:
Overall Officials: Richard Leigh, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share IPD with other researchers